CLINICAL TRIAL: NCT06933342
Title: Evaluating an Integrated Habituation Programme for Enhancing Dental Examination Acceptance in Children With Autism Spectrum Disorder: An Effectiveness Trial
Brief Title: ASD and Habituation to Dental Examination
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oral Health Center of Expertise Rogaland, Norway (Other)
Collaborators: University of Oslo (Other); The public dental health service Vestland Norway (Unknown); Oral Health Centre of Expertise in Western Norway (Other); The public dental health service Rogaland Norway (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OralHealthRogaland
Record Dates: First submitted 2025-03-10; First posted 2025-04-18 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Oral Health Training; Habituation; Autism Spectrum Disorder
Keywords: autism spectrum disorder; ASD; Dental examination; Dental habituation programme; Habituation; Oral health training
MeSH Terms: conditions — Substance-Related Disorders; Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: A pragmatic randomized controlled trial will be employed to assess the effectiveness of a habituation program for children with autism spectrum disorders to enhance cooperation between the child and the dental hygienist and to enable a dental examination at a local dental clinic. Children will be assigned to either a habituation group (five habituation sessions) or to a control group receiving a "toolbox" with visual aids for preaparations at home.
Who Masked: Outcomes Assessor
Masking Description: To investigate the effectiveness of the intervention (the habituation program), blinded dental personell (not part of the study otherwise) will perform an oral examination (treatment as usual) on the children approx. 6 weeks following the first habituation/starting preparation at home.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- At home preparation (Other): The control group will be an augmented control group. The participants in this group will receive a "toolbox" with visual aids and a dental examination mirror and written instructions on how to use the toolbox for preparations at home prior to the dental appointment
  Interventions: Behavioral: Preparations at home
- Habituation group (Experimental): Participants in the experimental group will receive five structured habituation sessions in a dental clinic with a trained dental hygienist. Parents/guardians will receive a "toolbox" with visual aids, a dental examination mirror and instructions for use at home preparations prior to the habituation sessions.
  Interventions: Behavioral: Habituation to dental examination

INTERVENTIONS:
Behavioral: Habituation to dental examination — The habituation will be performed by dental hygenists working in the public dental service in Rogaland or Vestland counties. The dental hygenists have completed a 2-day educational course consisting of both theoretical and practical information specifically adressing dental examination of children with autism spectrum disorder. The habituation will be done at the dental office.
  The intervention consists of five structured habituation sessions with the trained dental hygienist where the different elements of a clinical dental examination will be introduced stepwise in a controlled manner. Parents/guardians will also receive a "toolbox" with visual aids and a dental examination mirror with instructions for use during home preparations prior to the habituation sessions.
  Arms: Habituation group
Behavioral: Preparations at home — Participants in the augmented control group will receive a "toolbox" with visual aids and a dental examination mirror. The parents/guardians of these participants will receive written information on how to use these tools at home to prepare for a clinical dental examination.
  Arms: At home preparation

SUMMARY:
The goal of this effectiveness trial is to investigate if an integrated dental habituation programme can enhance acceptance of a clinical dental examination in children (aged 5-8 years) with autism spectrum disorder (ASD).

The main questions it aims to answer are:

* Can a dental habituation programme performed by trained dental hygienists increase the acceptance of a clinical dental examination in children with ASD?
* Is a dental habituation programme for children with ASD more effective compared to home preparation using visual aids performed by parents/guardians in increasing the acceptance of a clinical dental examination in children with ASD?

The study participants will be randomly assigned to either the habituation group (intervention) or the home preparation group (augmented control) to investigate the effectiveness in increasing acceptance and cooperation of a clinical dental examination.

DETAILED DESCRIPTION:
BACKGROUND Autism Spectrum Disorder (ASD) is a developmental disorder characterized by deviations in language, communication, social interaction, and a restricted and repetitive pattern of activities and interests. Good oral health is crucial for life satisfaction and impacts general health, nutrition, appearance, and communication. Several studies have shown that children with ASD often face challenges during oral examinations and dental treatments. Increased stress and anxiety in these patients also make dental treatment challenging for caregivers and the dental team. Various studies have demonstrated that communication aids, such as visual tools (pictures, books, films), and familiarization techniques (e.g., tell-show-do), can reduce stress and increase cooperation during dental examinations. Studies indicate that knowledge about ASD among healthcare professionals is limited. Despite continuous improvements, there is significant variation in knowledge levels across different age groups and professional backgrounds. A lack of knowledge and confidence in their skills among healthcare professionals can result in poorer healthcare services for children with ASD. Sufficient knowledge and early intervention are essential for achieving positive outcomes for this patient group.

METHODS

Design and Procedures:

To address this challenge and enable more dental examinations at local clinics, the investigators have developed a training program for dental personnel. The course, developed by pediatric dentists, was presented to a resource group consisting of a psychologist, a dental hygienist, dentists, a researcher, and a parent of a child with ASD. Adaptations were made based on feedback from the resource group. The course includes both theoretical and practical content, focusing on ASD characteristics, communication techniques, and tools specific to this patient group to increase cooperation and the completion of clinical dental examinations. During the course, dental personnel will be trained in a habituation program to provide a gradual and structured approach to dental examinations, minimizing unwanted behavior and reducing perceived stress in the child, parent, and dental practitioner. To the effectiveness of the integrated habituation program will be evaluated in a randomized controlled trial. The intervention will last for 5 weeks, with one habituation session each week. The habituation sessions will be performed at selected dental clinics. Clinics will be selected based on geographical location, and on the affiliation of the dental hygienist participating in the study.

Participants will be recruited from two counties in western Norway (Rogaland and Vestland) and randomly assigned to either the intervention group or an augmented control group. The augmented control group will receive a toolbox with visual aids for home preparation before a dental appointment, similar to the intervention group. Participation will be based on written informed consent provided by the parents og caregivers of the children.

Measurements:

The effects of the habituation program will be assessed based on the successful completion of a clinical dental examination. Additionally, changes in cooperation (using the Frankl scale) during each session will be recorded. Parents will be asked to fill out a mapping form at baseline, and clinical data from patient journals will be collected. Child stress will be measured using the Wong Baker FACES® scale. In addition, following the intervention, both parents and dental hygieneists will be invited to an interview to share their experiences as part of the evaluation of the study.

Power and Sample Size:

The estimation of sample size is based on a binary logistic model with a random effect factor. 1000 Monte Carlo simulations indicate that 225 children are needed to provide satisfactory power, given that the difference in the probability of success is not less than 0.2. However, there is uncertainty associated with the calculations since previous studies, which formed the basis for this calculation, differ from this study in several ways (e.g., different age and setting, different steps in the habituation program). It was calculated that at least 6 dental hygienists are needed to participate in the study and perform the habituation program.

Data Analysis:

The statistical software package SPSS (IBM) will be used to analyze quantitative data such as questionaire data, Frankl scale data, and clinical data from patient journals. The analyses will include descriptive statistics and statistical tests to identify changes and differences in the study variables within and between the intervention and control groups (e.g., t-tests, mixed-effects models). It is hypothesized that the use of the habituation program will lead to increased cooperation and completion of clinical dental examinations, and a reduction in child and parental stress in this setting. Regression analysis will be employed to investigate associations between study variables while adjusting for potential covariates. NVivo (Alfasoft) will be used to analyze additional qualitative data from patient journals.

ELIGIBILITY:
Inclusion Criteria:

* Children living in the counties Rogaland or Vestland, Norway
* English or Norwegian speaking
* Have not been able to complete a clinical dental examination at the local dental clinic
* Has an autism spectrum diagnosis (reported by parents/guardians)

Exclusion Criteria:

* Children not living in the counties Rogaland or Vestland, Norway
* Does not speak English or Norwegian
* Have completed a dental examination at the local dental clinic
* Have other severe developmental cognitive disabilites (in addition to an autism spectrum diagnosis) (reported by parents/guardians)

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 225 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Completion of a clinical dental examination with good cooperation | 6 weeks after the first habituation session/home preparation
  The dental examination has been divided into several steps (i.e., sitting in the chair, accepting examination with dental mirror, accepting light from the lamp, examination with probe). The primary objective will be completion of a clinical dental examination (examination with mirror and probe) with good cooperation. After 5 weeks (either with home preparation or habituation sessions) a blinded dental personell (untrained) will do a clinical dental examination (treatment as usual). Cooperation will be measured using the Frankl scale, reported by the parents/guardians for each step in the dental examination.

SECONDARY OUTCOMES:
Changes in child stress measured by Wong-Baker FACES pain rating scale | At session 1, (only intervention group), after 6 weeks (intervention and control group)
  Changes in child stress will be measured by Wong-Baker FACES pain rating scale. The children will be asked to indicate how they feel by pointing on one of the faces that best describe how they feel. If the child is not capable of performing this task, the parent/guardian will be asked to indicate on the scale how they perceive their child to feel at that moment. Children in the intervention group will be asked to do this at the first habituation session and at the post-test (approx. 6 weeks later). Children in the control group will only perform the rating once, at the post-test.
Changes in cooperation assessed by Frankl scale | Once per week for 5 weeks
  For the intervention group, cooperation during each habituation sessions will be monitored using the Frankl scale. Parents/guardians will be asked to fill out the form.

OTHER OUTCOMES:
Mapping questionnaire | Day 0
  At enrollment, parents/guardians will be asked to fill out a questionnaire mapping age, gender, communication skills, sensitivites, previous experience with the public dental service, behavior, oral hygiene habits.
Oral health status measured by DMFT | Day 0
  To map the oral status of the children and potential unmet needs DMFT will be collected from the patient records. Data collection will be performed by dental personnel with access to the patient record system (OPUS).
Oral hygiene measured by BSI or equivalent measurement | At the last habituation session (session 5), week 5
  To map the hygiene of the children, BSI will be assessed either during the last habituation session, if possible, or otherwise collected from the patient records. Data collection will be performed by dental personnel with access to the patient record system (OPUS).
Interview with dental hygienist's to gain their experiences with participating in the study | Periprocedural, within 2-3 months
  As part of evaluating the effectiveness of the study and the implementation into a regular dental practice, the dental hygienists who performed the habituation sessions will be interviewed. Their feedback will be important for the future development of the habituation programme and enable the incorporation of the habituation programme into the public dental service. Interviews will be semi-structured focusing on their experiences, motivation for participation, potential or experienced barriers or success factors, development of the habituation programme, implementation
Interveiw with parent's to evaluate the study (habituation programme and home training) | Periprocedural, within 2-3 months
  To gain insight into the effectiveness of the study and get the user perspective, parents will be interviewed after completion of the intervention. Their answers could inform the future development of the habituation programme and the "toolbox". The interviews will follow a semi-structured interview guide focusing on their experiences with participating in the study. Parents will be invited to participate in an interview (by telephone or video conference call) after the intervention is finished.

CONTACTS AND LOCATIONS:
Overall Officials: Lene Elisabeth Myhren, PhD, Principal Investigator — Oral health centre of expertise - Rogaland, Norway
Locations (2):
- Norway (2):
  - Oral health centre of Expertise Rogaland, Stavanger, Rogaland
  - The public dental health service Vestland Norway, Bergen, Vestland

IPD SHARING:
Plan to Share IPD: No
IPD from this study will not be shared with researchers outside the project group. This is emphasized in the information- and consent form that iwll be handed out to the participants (their parents/guardians) prior to data collection.